CLINICAL TRIAL: NCT04372056
Title: A Norwegian Study on Views and Experiences of Health Care Professionals Working in Intensive Care Units During the COVID-19 Pandemic.
Brief Title: The COVID-ICU Healthcare Professional Study
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Irene Lie, Principal investigator, RN, CCN,PhD, Oslo University Hospital
Other Study IDs: 136144
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: COVID-19; Critical Care; Intensive Care Units; Health Personnel
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Views and experiences of health care professionals working in intensive care units during the COVID-19 pandemic — Health care professionals
  Other Names: COVID-ICU Health Care Professionals

SUMMARY:
The project is a longitudinal cohort study based on an electronic questionnaire on views and experiences of COVID-ICU Health care professionals during the pandemic. In addition, a few of the informants participating in the cohort study will be asked to participate in focus groups to get a deeper understanding of the experiences of Health care professionals. Leaders at the randomized hospitals will be asked to participate in individualized interviews.

DETAILED DESCRIPTION:
Health Care professionals in intensive care units (ICU) are working front-line with coronavirus disease (COVID-19) patients with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in need of intensive care treatment.

Data collected will identify the health care professionals' (nurses, medical doctors, leaders) views and experiences from the planning period of COVID-19 ICU units until a follow-up at 12 months.Themes to be covered in the survey are organization, information, communication across disciplines, education, practical implementation, use of personal protective equipment, daily working conditions and psychosocial aspects. The Oslo University Hospital/University of Oslo, GDPR (General Data Protection Regulation) compliant "TSD"-Services for Sensitive data web-based solution "Nettskjema" will be used combined for consent form and data collection from the survey. It is within the scope of the study to perform sub analysis on background variables as profession related to daily working experiences on COVID-ICU and psychosocial aspects.

A few of the informants (medical doctors, nurses, leaders) participating in the cohort study will randomly (computerized) be asked to participate in focus groups to get a deeper understanding of the experiences of the health care professionals during the pandemic and after the pandemic when they are back to a normal working condition. Leaders at the randomized hospitals will be asked to participate in individualized interviews. Data from the focus group interviews and individual interviews will be taped on a recorder approved by data protection officer at Oslo University Hospital and then stored at a secured computerized research place at Oslo University Hospital.

The gained knowledge from both the survey, the focus group interviews and individual interviews in this study may guide hospital directors and the government in follow up of health care professionals and to prepare for a later pandemic.

ELIGIBILITY:
Inclusion Criteria:

All health care professionals (nurses, medical doctors, leaders) working in all COVID-ICUs in Norway will be invited to participate in this project.

Exclusion Criteria:

No exclusion criteria

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The longitudinal cohort study will collect data from all consenting health care professionals in COVID-ICUs in Norway during the pandemic with 3- and 12-months follow-up on a combined electronic consent form and questionnaire that the informants will fill in using a computer and an electronic identification.
  A few of the informants (medical doctors, nurses, leaders) participating in the cohort study will randomly (computerized) be asked to participate in focus groups during the 12-months study follow-up. Leaders at the randomized hospitals will be asked to participate in individualized interviews.
Sampling Method: Non-Probability Sample
Enrollment: 484 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Views and experiences of health care professionals working in intensive care units during the COVID-19 pandemic | 1 year
  Health care professionals working in COVID-ICUs

CONTACTS AND LOCATIONS:
Overall Officials: Irene Lie, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo university hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hovland IS, Skogstad L, Stafseth S, Hem E, Diep LM, Raeder J, Ekeberg O, Lie I. Prevalence of psychological distress in nurses, physicians and leaders working in intensive care units during the COVID-19 pandemic: a national one-year follow-up study. BMJ Open. 2023 Dec 22;13(12):e075190. doi: 10.1136/bmjopen-2023-075190. PMID 38135308
- [Derived] Lie I, Stafseth S, Skogstad L, Hovland IS, Hovde H, Ekeberg O, Raeder J. Healthcare professionals in COVID-19-intensive care units in Norway: preparedness and working conditions: a cohort study. BMJ Open. 2021 Oct 11;11(10):e049135. doi: 10.1136/bmjopen-2021-049135. PMID 34635518